CLINICAL TRIAL: NCT00138138
Title: Psychostimulants for Fatigue in Advanced Prostate Cancer
Brief Title: Psychostimulants for Fatigue in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fordham University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-100
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Fatigue; Prostate Cancer
MeSH Terms: conditions — Fatigue; Prostatic Neoplasms | interventions — Methylphenidate

INTERVENTIONS:
Drug: Ritalin

SUMMARY:
Fatigue is one of the most common symptoms of prostate cancer. Fatigue is a lack of energy that makes it harder to do the things you normally do every day. Some symptoms of fatigue are:

* feeling tired and/or weak;
* having less interest in activities;
* having trouble concentrating;
* feeling "down";
* feeling exhausted for no clear reason.

There are not many drugs that are helpful in treating fatigue. However, one group of medications does seem to be useful. In this study, we, the investigators at Memorial Sloan-Kettering Cancer Center, will be using a psychostimulant called Ritalin. The aim of this study is to see if this drug is helpful in treating fatigue in prostate cancer. We are also studying the side effects of this medication.

DETAILED DESCRIPTION:
This study is open to men who have prostate cancer and report feeling fatigue. We will examine the impact of psychostimulant treatment on depressive symptom severity, neuropsychological test performance, and overall quality of life, as well as compare the frequency and severity of treatment associated adverse side effects. We will be conducting a six-week, randomized, double-blind, placebo-controlled, parallel design trial, evaluating the relative benefits and risks of methylphenidate, (a psychostimulant medication). Medication will be given in once or twice daily dosages (at 8 am and noon) and titrated by one capsule every 2-3 days as needed to treat fatigue and as tolerated. Patients will be examined regularly for safety. We will monitor vital signs and response to the medication. This study will be the first of its kind to evaluate a pharmacologic intervention for fatigue in cancer patients that utilizes a novel psychotropic agent (psychostimulant), and assesses outcome with measures of fatigue, as well as side effects, psychological distress, depression and overall quality of life.

Objectives: To study the efficacy of methylphenidate vs. placebo in the treatment of fatigue in ambulatory men with prostate cancer.

To study the frequency and severity of adverse side effects associated with this psychostimulant drug.

To study the effects of psychostimulant treatment for fatigue on related domains of psychosocial function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and English speaking (patients who cannot read will be offered assistance with the consent forms and surveys). There is no maximum age cut off for eligibility into this study.
* Diagnosed with prostate cancer.
* Receiving ambulatory medical care at the time of initial assessment and primary treating physician is aware of and agrees to the subject's participation in the study.
* Fatigue that has been persistent (chronic-recurrent or continuous for a period of at least 2 weeks), and is reported to have an intensity of moderate or severe (a score of 4 or greater on one question that assesses fatigue over a two week period on a 0-10 numeric rating scale).
* Patients who have already received six weeks of Procrit therapy at 60,000 units for anemia and still have significant fatigue will then become eligible for this stimulant trial.
* Patients who have received three weeks of thyroid supplementation therapy for hypothyroidism and still have significant fatigue will then become eligible for this stimulant trial.
* Patients who are able to give informed consent.

Exclusion Criteria:

* Significant cognitive impairment (Mini-Mental Status score of 22 or below) or psychiatric disturbance sufficient, in the investigator's judgment, to preclude data collection and informed consent.
* Evidence of severe renal or hepatic disease; serum creatinine and liver function tests (LFT's) must be no higher than 2 times the upper limit of normal.
* A white blood cell count below 2,000 cells per cubic millimeter or platelets 60,000 per cubic millimeter or less.
* Uncontrolled hypertension (blood pressure [BP] of 170/100 or greater) will exclude patients from the study. For those patients with histories of controlled hypertension (either by diet or medication), methylphenidate may increase resting blood pressure by 5 mmHg. (The patients will have blood pressure, pulse and other vital signs monitored weekly under the auspices of the Genitourinary Clinic, or at home under the instruction of the research nurse, using a blood pressure monitor issued by the study.)
* Urgent need of a primary medical therapy for fatigue that would be more appropriate than the study drug (eg, severe anemia where the hemoglobin is less than 11.0 or if the patient is symptomatic. Patients who have already received six weeks of Procrit therapy and still have significant fatigue will then become eligible for this trial).
* Patients found to have significant hypothyroidism (as defined by thyroid stimulating hormone test greater than 4.42 upon blood chemistry screening), will be ineligible for this study until they have completed three weeks of appropriate thyroid supplementation and are still found to exhibit significant fatigue.
* History of substance abuse (ie, stimulant drugs, cocaine, or injection drug use) or participation in a methadone maintenance program. Patients with a history of alcohol abuse will not be excluded from this study if they are currently not abusing alcohol.
* Meeting criteria for a diagnosis of major depressive episode - current (screening for major depression will be completed using the Structured Clinical Interview for DSM-IIIR, Nonpatient Version [SCID-NP]). Concurrent use of monoamine oxidase (MAO) inhibitors, tricyclic antidepressants, or a psychostimulant will exclude subjects from study participation. Concurrent use of other antidepressant medications (eg, selective serotonin reuptake inhibitors [SSRIs], serotonin-norepinephrine reuptake inhibitors [SNRIs]) will not exclude subjects from study participation.
* History of allergy to, or intolerance of, methylphenidate.
* Karnofsky Patient Performance Rating score of 50 or below.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-10; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To study the efficacy of methylphenidate (Ritalin) versus placebo in the treatment of fatigue in ambulatory men with prostate cancer

SECONDARY OUTCOMES:
To study the frequency and severity of adverse side effects associated with this psychostimulant drug
To study the effects of psychostimulant treatment for fatigue on related domains of psychosocial function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Roth, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org